CLINICAL TRIAL: NCT03174262
Title: Effects of an Occupational Therapy Computer Workstation Intervention on Ergonomic Knowledge, Self-efficacy, and Habit Formation
Brief Title: Effects of an OT Workstation Intervention on Knowledge, Self-efficacy, and Habit Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HM20006719
Record Dates: First submitted 2017-04-21; First posted 2017-06-02 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Occupational Injuries
Keywords: Ergonomics; Computer Workstation; Habit; Self-efficacy; Knowledge
MeSH Terms: conditions — Occupational Injuries; Habits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ergonomic Computer Workstation Training (Experimental)
  Interventions: Behavioral: Ergonomic Computer Workstation Training
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Ergonomic Computer Workstation Training — Training in proper body alignment and use of computer at computer workstations for people who spend 30% or more of a typical day at a computer. Training consists of learning proper positioning for head, neck, shoulders, arms, hands, and legs; proper arrangement of computer monitor, keyboard, mouse, and accessories.
  Arms: Ergonomic Computer Workstation Training

SUMMARY:
The study aims to determine whether a face to face ergonomic workstation intervention has any advantage over an online instructional training program for acquisition of knowledge, self-efficacy, and habit formation.

DETAILED DESCRIPTION:
Thirty participants will be recruited from the staff of Virginia Commonwealth University via recruitment fliers distributed through the Staff Senate. Potential participants will be informed that participation in the study will require them to work with the research team at their computer workstations outside of designated working hours, e.g., before or after work, during lunch break, or on a weekend. Potential participants will be reminded that they may need to obtain approval from direct supervisors to use university equipment, i.e., their computer workstations, during non-working hours. All participants will be asked to complete knowledge, self-efficacy, and habit formation survey regarding computer workstation ergonomics via REDCap.

Participants will receive an email with the link to the REDCap surveys.

Those participants randomly assigned to the control group will complete the OSHA Computer Workstations eTool, available at (https://www.osha.gov/SLTC/etools/computerworkstations/wkstation_enviro.html). The eTool consists of 5 sections: 1) Good Working Positions, 2) Workstation Components, 3) Checklists, 4) Work Process, and 5) Workstation Environment.

Those participants who are assigned to the intervention group will be contacted by the investigators to schedule face to face visits at their computer workstations. Face to face intervention will consist of educating the participant on points of computer workstation ergonomics, direct observation of the participant working at her/his workstation, evaluation of workstation characteristics, instruction on how to alter workstation features, and instruction on best practices for exercise and scheduling of breaks to prevent pain, discomfort, and injury.

All participants will be contacted via email 2 weeks following the interventions to complete the post-test knowledge, self-efficacy, and habit formation survey on RedCap.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old or older.
* Work at computer workstation at least 30% of a typical day.

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Change in Knowledge, Self-efficacy, and Habit Formation Survey score | Pre- and Two Weeks Post-Intervention
  Aggregate score from survey

CONTACTS AND LOCATIONS:
Overall Officials: Al Copolillo, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers.